CLINICAL TRIAL: NCT05721508
Title: Effect of Practice Environment on Perceived Benefits of Combined Physical and Cognitive Program on Older People's Cognitive Abilities and Quality of Life
Brief Title: Cognitive and Physical Stimulation and Promotion of Social Relations for the Benefit of Older People's Quality of Life
Acronym: StimCoAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Poitiers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAPR2021-2020-12021410
Record Dates: First submitted 2023-01-17; First posted 2023-02-10 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Aging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Individual practice at home (Experimental): Participants will undergo a training program combining physical and cognitive activities in individual practice at home.
  Interventions: Other: Combined physical and cognitive program
- Group practice in a traditional group environment (gymnasium) (Experimental): Participants will undergo a training program combining physical and cognitive activities in group practice in a traditional group environment (gymnasium).
  Interventions: Other: Combined physical and cognitive program
- Group practice in an enriched environment fostering social relations (Experimental): Participants will undergo a training program combining physical and cognitive activities in group practice in an enriched environment fostering social relations.
  Interventions: Other: Combined physical and cognitive program

INTERVENTIONS:
Other: Combined physical and cognitive program — All participants will complete 12-week training sessions combining physical and cognitive activities, with two 1-hour sessions per week.

SUMMARY:
The aim of this interventional study is thus to assess and highlight the cognitive, physical, and psychosocial benefits of a combined physical and cognitive training program in an enriched environment and to assess the factors influencing these benefits.

DETAILED DESCRIPTION:
The number of older people worldwide is constantly increasing. However, one of the main problems associated with aging is cognitive decline, which affects essential everyday functions such as memory, attention, and executive functions. Thus, maintaining autonomy and quality of life depends on physical health, and the integrity of cognitive functioning. Cognitive, physical and social activities can all slow this decline but social factors and their contribution to the well-being of older people remain under-researched. The aim of the present study is to analyze how the practice environment can foster these social relations and thus enhance wellbeing and to identify the psychological dimensions that are activated by social relations.

ELIGIBILITY:
Inclusion Criteria:

* People must be at least 65 years old
* People must be at independent (able to get around on their own: car, bus, walking)
* People must be at living in the community (not in an institution such as a nursing home)
* The persons recruited must have a score on the Montreal Cognitive Assessment (MoCA) of at least 18.

Exclusion Criteria:

* People with contraindications for engaging in regular physical activity
* People with severe neurological and psychological disorders.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 172 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2024-12-20 (Actual); Study Completion 2024-12-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline Score at Trail Making Test (TMT) | inclusion; 6 weeks; 12weeks; 9 months
  Score at cognitive flexibility function. higher scores mean a worse outcome.
Change from baseline Score at Stroop task | inclusion; 6 weeks; 12weeks; 9 months
  Score at cognitive inhibition function. higher scores mean a worse outcome.
Change from baseline Score at N-Back task | inclusion; 6 weeks; 12weeks; 9 months
  Score at working memory updating. Higher scores mean a better outcome
Change from baseline Score at Montreal Cognitive Assessment (MoCA) | inclusion; 6 weeks; 12weeks; 9 months
  Score at basic cognitive functions. Higher scores mean a better outcome
Change from baseline Score at letter comparison test (XO test) | inclusion; 6 weeks; 12weeks; 9 months
  Score at processing-speed of information. Higher scores mean a better outcome
Change from baseline Score at Remember-Know paradigm | inclusion; 6 weeks; 12weeks; 9 months
  Score at episodic memory. Higher scores mean a better outcome
Change from baseline Score at 16-item Free and Cued Recall | inclusion; 6 weeks; 12weeks; 9 months
  Score at episodic memory. Higher scores mean a better outcome
Score at Mill-Hill vocabulary test | Inclusion
  Score at crystallized intelligence. Higher scores mean a better outcome
Change from baseline Score at Social Provisions Scale [SPS-10; score: 10-40]. (self-report questionnaire) | inclusion; 6 weeks; 12weeks; 9 months
  Perceived social support Score (attachment, social integration, confirmation of one's value, material help, orientation) (self-assessment). Higher scores mean a better outcome.
Change from baseline Score at Rosenberg's Self-Esteem Scale [EES-10; score: 10-40] (self-report questionnaire) | inclusion; 6 weeks; 12weeks; 9 months
  Perceived self-esteem Score (self-assessment). Higher scores mean a better outcome.
Change from baseline Score at French Achievement Goals Questionnaire for Sport and Exercise (QFBASEP) (self-report questionnaire) | inclusion; 6 weeks; 12weeks; 9 months
  Goal of motivation for physical activity (self-assessment)
Change from baseline Score at 5-item World Health Organization well-being index [WHO-5; score: 0-100] (self-report questionnaire) | inclusion; 6 weeks; 12weeks; 9 months
  Perceived well-being Score (self-assessment). Higher scores mean a better outcome.
Change from baseline Score at Mental Health Continuum Short Form [MHC-SF; score: 0-70] (self-report questionnaire) | inclusion; 6 weeks; 12weeks; 9 months
  Perceived emotional, social and psychological well-being Score (self-assessment). Higher scores mean a better outcome.
Change from baseline Score at anxiety item on Hospital Anxiety and Depression Scale [HADS; score: 0-21] (self-report questionnaire) | inclusion; 6 weeks; 12weeks; 9 months
  Anxiety Score (self-assessment). higher scores mean a worse outcome.
Change from baseline Score at depression item on Hospital Anxiety and Depression Scale [HADS; score: 0-21] (self-report questionnaire) | inclusion; 6 weeks; 12weeks; 9 months
  Depression Score (self-assessment). higher scores mean a worse outcome.
Semi-structured interview | inclusion; 6 weeks; 12weeks; 9 months
  Assessment of social and cultural life, and assessment of interactions and relations with group members or teachers: "How would you describe your social and cultural life now?", "How the sessions with the other members of the group going?"
Change from baseline Score at level of physical activity and sedentary lifestyle questionnaire (ONAPS) | inclusion; 6 weeks; 12weeks; 9 months
  Level of physical activity and sedentary lifestyle
Change from baseline Score at Dynamic balance and walking speed with Time Up and Go test | inclusion; 6 weeks; 12weeks; 9 months
  Dynamic balance and walking speed. A shorter time means a better result
Change from baseline Score at 30-second Chair Stand Test | inclusion; 6 weeks; 12weeks; 9 months
  Score at lower body strength. Higher scores mean a better outcome
Change from baseline Score at arm Curl Test | inclusion; 6 weeks; 12weeks; 9 months
  Score at upper body strength. Higher scores mean a better outcome
Change from baseline Score at six Minutes' Walk Test (6MWT) | inclusion; 6 weeks; 12weeks; 9 months
  Aerobic capacity. Higher distance traveled means a better result

CONTACTS AND LOCATIONS:
Overall Officials: David Clarys, Study Director — University of Poitiers
Locations (1):
- University of Poitiers, Poitiers, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gonnord T, Clarys D; StimCoAPS Consortium; Dupuy O, Albouy M, Migeot V, Grangeiro R, Esnard C, Boucard G. Effects of combined physical and cognitive program performed in socially enriched environment on older people's cognitive abilities and quality of life (StimCoAPS): study protocol for a randomized controlled trial. BMJ Open Sport Exerc Med. 2023 Oct 11;9(4):e001577. doi: 10.1136/bmjsem-2023-001577. eCollection 2023. PMID 37860154